CLINICAL TRIAL: NCT04846270
Title: An Open, Single-arm, Post-market Clinical Investigation to Verify the Ability of TENA SmartCare Change Indicator to Reduce the Number of Manual Checks Between Changes of Absorbing Incontinence Products in a Home Environment.
Brief Title: Investigation of the Ability of the TENA SmartCare Change Indicator to Reduce the Number of Manual Checks Between Changes of Absorbing Incontinence Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: POWER
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2023-10

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Device (Experimental): TENA SmartCare Change Indicator
  Interventions: Device: TENA SmartCare Change Indicator

INTERVENTIONS:
Device: TENA SmartCare Change Indicator — Each participating subject will be provided with TENA SmartCare Change Indicator and incontinence products for the duration of the investigation. Each participating subject will be allocated to the incontinence type(s) that are considered most suitable.

SUMMARY:
The purpose of this post market clinical investigation is to demonstrate the performance and safety of the TENA SmartCare Change Indicator.

DETAILED DESCRIPTION:
The TENA SmartCare Change Indicator is intended for use on individuals, dependent end user (DEU), suffering from Urinary Incontinence (UI) who are cared for in a home environment, by one or more caregivers (CGR). The TENA SmartCare Change Indicator is an accessory to TENA absorbing incontinence products. This clinical investigation is intended to demonstrate that use of TENA SmartCare Change Indicator has the ability to reduce the number of manual checks between daily changes of absorbing incontinence products. Secondarily, the investigation will evaluate number of leakages, skin redness, usability and fecal incidence. Furthermore, the safety will continuously be monitored through analyzing device-related adverse events reported during the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. DEU is diagnosed with urinary incontinence managed with a tape-style incontinence product.
2. DEU is unable to sufficiently communicate the need for an incontinence product to be changed.
3. DEU is being cared for in a home environment and most of the care is provided by a main CGR.
4. DEU is willing and able to provide informed consent and to participate in the clinical investigation or has a legally designated representative willing to provide informed consent on behalf of the DEU. Note, the legally designated representative and main CGR cannot be the same person.
5. CGR is willing and able to provide informed consent to participate in the clinical investigation.
6. The CGR frequently checks the saturation level of the incontinence product, manually and/or by a touch-feel process.
7. If incontinence is managed by pharmaceuticals, the dose regime is stable.
8. DEU and CGR ≥ 18 years of age.

Exclusion Criteria:

1. DEU is cared for in a professional establishment or is institutionalized.
2. DEU has ≥ 4 fecal "incidences" per week.
3. DEU has severe incontinence product related skin problems, as judged by the investigator.
4. DEU has any type of urinary catheter(s) resulting in improved/treated urinary incontinence.
5. The incontinence product is changed on a routine based on time (schedule) or device alert, without manual checks.
6. Any other condition that may make participation in the clinical investigation inappropriate, as judged by investigator.
7. CGR is incapable or unwilling to use the required smart phone application and/or the diary registration webpage required for the clinical investigation.
8. Participation in an investigational study of a drug, biologic, or device within 30 days prior to entering the clinical investigation or planned during the course of the clinical investigation.
9. DEU is pregnant or nursing.
10. CGR or DEU with an alcohol or drug addiction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Piotr Radziszewski, MD, PhD, Principal Investigator — Medical Concierge Centrum Medyczne, Polnej Rózy 6/U2, 02-798 Warszawa,
Locations (1):
- Medical Concierge Centrum Medyczne, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Device
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 35
General Cognitive Function [Number; unit: participants] — The principal investigator general assessment of the cognitive function of the participant i.e if there are any confusion or dementia present.
  participants
    No cognitive impairment | 5
    Mild cognitive impairment | 26
    Severe cognitive impairment | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Manual Checks Per Day at Baseline Week and 3 Weeks
Description: A comparison between the average number of manual checks, in-between the regular changes of the absorbing incontinence product, in the third week of the study (investigational week) and the first week of the study (baseline week).
Time Frame: 3 weeks
Population: The population consist of all consented subjects that do not have a major protocol deviation and have at least one set of efficacy measurements after using the investigational device
Measure: Mean (Standard Deviation); unit: Checks per day
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
Checks per day
  Investigational week | 3.5 (2.0)
  Baseline week | 4.3 (1.8)
Statistical Analysis 1: Comparison: Investigational Device; POWER is a single arm investigation with cross-over design. Each participating subject will use the study device and act as its own control. The null hypothesis (H0) is that there is no difference in the mean number of checks performed during the investigation week compared to the baseline week. The alternate hypothesis (H1) is that there is a reduction in the mean number of checks performed during the investigation week compared to the baseline week; Test type: Other; p = 0.0006, Wilcoxon (Mann-Whitney); A Wilcoxon Signed-Rank test was used to test if the number of manual checks has been reduced

2. Secondary Outcome: Number of Safety Related Events
Description: Reported number of adverse events (AE), adverse device effects (ADE), serious adverse events (SAE), serious adverse device effects (SADE), and device deficiency (DD) as reported in the investigation.
Time Frame: 3 weeks
Population: The population consist of all consented subjects.
Measure: Number; unit: Occurences
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
Occurences
  Adverse events | 5
  Adverse device effects | 0
  Serious adverse events | 0
  Serious adverse device effects | 0
  Device deficiency | 39

3. Secondary Outcome: Number of Leakages Per Day Into the Clothes and/or Bed Linen at Baseline and 3 Weeks
Description: A comparison between the average number of urine leakages (out of the absorbing incontinence product), onto the clothes and/or bed linen, in the third week of the study (investigational week) and the first week of the study (baseline week).
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Leakages per day
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
Leakages per day
  Investigational week | 0.2 (0.37)
  Baseline week | 0.33 (0.44)
Statistical Analysis 1: Comparison: Investigational Device; Test type: Other; p = 0.0051, Wilcoxon (Mann-Whitney); A Wilcoxon Signed-Rank test was used to test if the number of leakages had been reduced

4. Secondary Outcome: Number of Participants With Skin Redness and Irritation
Description: A comparison between investigational (week 3) week and baseline week (week 1). The Ghent Global IAD Categorisation Tool (GlOBIAD) was used. It has a 4 point scale from minimum 1A to maximum 2B (with 1A being better outcome). In the measure. IAD is incontinence associated dermatitis.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
Participants
  Investigational week No visible skin redness or irritation. | 35
  Investigational week GLOBIAD score 1A | 0
  Investigational week GLOBIAD score 1B | 0
  Investigational week GLOBIAD score 2A | 0
  Investigational week GLOBIAD score 2B | 0
  Baseline week. GLOBIAD score 1A. | 2
  Baseline week. No visible skin redness or irritation. | 33
  Baseline week. GLOBIAD score 1B. | 0
  Baseline week. GLOBIAD score 2A. | 0
  Baseline week. GLOBIAD score 2B. | 0

5. Secondary Outcome: Usability Assessed Via Caregiver-reported Questions With a Qualitative Scale at the End of the Study.
Description: Average score is presented. The scale is 5-point, from minimum 1 to maximum 5 (with 5 being the better outcome).
Time Frame: At the end of investigational week (week 3).
Population: The population consist of all consented subjects that do not have a major protocol deviation and have at least one set of efficacy measurements after using the investigational device. For the questionnaire these questions were answered by the care giving relative.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
score on a scale
  How would you evaluate the written instructions for use of the system? | 4.7 (0.5)
  How easy was the Change Indicator to use? | 4.8 (0.5)
  How easy was the app to use? | 4.9 (0.3)
  How would you grade the overall usefulness of the system? | 4.4 (0.9)

6. Secondary Outcome: Number of Fecal Incidences.
Description: Presented in listing. No formal endpoint. Will only be used for assessing reliable primary endpoint measurements.
Time Frame: 3 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Fecal episodes per day
Arm/Group | Investigational Device
Number analyzed (Participants) | 35
Fecal episodes per day
  Investigational week | 0.059 (0.178)
  Baseline week | 0.066 (0.215)
Statistical Analysis 1: Comparison: Investigational Device; Test type: Other; p = 0.76, Wilcoxon (Mann-Whitney); A Wilcoxon Signed-Rank test was used to test if the number of fecal incidents had been reduced

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Investigational Device
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 4/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=35)
Diarrhea (Infections and infestations) | 1 (2)
Urinary bleeding (General disorders) | 1 (1) — Blood in urine with visible blood clots
Pneumonia (Infections and infestations) | 1 (1)
Slightly raised temperature (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT04846270/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT04846270/SAP_001.pdf